CLINICAL TRIAL: NCT05948865
Title: A Phase 1, Multicenter, Single Agent Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of CPO301, an EGFR-Targeting Antibody-Drug Conjugate, in Adult Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1 Study of CPO301 in Adult Patients With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Conjupro Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPO301-US-101
Record Dates: First submitted 2023-06-22; First posted 2023-07-17 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Cancer, Lung
Keywords: Cancer; Non-Small Cell Lung Cancer; Solid Tumors; Metastatic; Advanced
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A, Dose Escalation (Experimental): Participants receive escalating doses of CPO301 of 0.6 mg/kg, 1.8mg/kg, 3.6 mg/kg, 4.8 mg/kg, 6.4 mg/kg and 8 mg/kg administered by IVI every 3 weeks (Q3W), with 21 days as a treatment cycle.
  Interventions: Drug: CPO301
- Part B, Dose Expansion (Experimental): Participants receive CPO301 at the recommended phase 2 dose (RP2D) determined in Part A, administered by IVI every 3 weeks (Q3W), with 21 days as a treatment cycle.
  Interventions: Drug: CPO301

INTERVENTIONS:
Drug: CPO301 — Administered by intravenous injection
  Other Names: SYS6010

SUMMARY:
The goal of this clinical trial is to test CPO301, a type of drug called an antibody drug conjugate in adult patients with advanced or metastatic solid tumors.

The main questions it aims to answer are:

* To assess the safety and tolerability of CPO301 at increasing doses and determine the dose to be used in the second part of the study (Part A)
* To assess the safety and tolerability of CPO301 at the dose determined to be safe and tolerable in Part A in patients with Non-Small Cell Lung Cancer and potentially other tumor types (Part B)
* To evaluate how quickly CPO301 is metabolized by the body (pharmacokinetics or PK)
* To evaluate if antibodies to the study drug develop (immunogenicity)
* To evaluate preliminary efficacy to the drug
* To correlate preliminary efficacy with mutations in a biomarker called EGFR

Participants will:

* Provide written informed consent
* Undergo screening tests to ensure they are eligible for study treatment
* Attend all required study visits and receive CPO301 by intravenous injection every 3 weeks until the study doctor determines study treatment should be stopped, based on how well a participant is doing on treatment
* Be followed for progression every 3 months for up to 2 years

DETAILED DESCRIPTION:
This Phase 1 study is a multicenter, dose-escalating, dose-expansion, single agent, 2-part study conducted in patients with advanced or metastatic solid tumors who progressed on ≥1 prior conventional systemic therapy or who were ineligible or intolerant to standard treatment or had no or refused standard treatment.

Dose escalation (Part A) - Dose escalation will be guided by a modified 3+3 design to determine the maximum tolerated dose (MTD) or recommended dose of CPO301 (also known as SYS6010). Determination of dose-limiting toxicity (DLT) will be based on toxicity observed during the DLT observation period (first 21 days [1 cycle]). Dose escalation decisions are made based on the occurrence of DLT. MTD will be determined based on the data of all enrolled participants. To better identify the MTD, one or more dose groups may also be added beyond the planned maximum dose group (if determined to be safe), or between the maximum escalation dose group and the next lower dose group for DLT assessment. Intermediate dose groups and/or adjustment to the dosing frequency may be made

Dose expansion (Part B) - Additional patients will be enrolled at the recommended dose determined in the dose escalation stage. An additional tumor cohort may be added based on data observed in Part A.

ELIGIBILITY:
Major Inclusion Criteria:

* Age ≥18 years
* Patients with histologically confirmed locally advanced or metastatic solid tumors who have disease progression, intolerance to prior therapy, are ineligible for available therapies, or refuse standard of care therapy in the metastatic setting.
* In Part A, patients with solid tumors including but not limited to NSCLC (adenocarcinoma and squamous cell carcinoma), breast cancer, KRAS-wild type colorectal cancer, and head & neck cancer based on previous biopsy result.
* In Part B, Cohort 1 will exclusively include NSCLC patients with documented EGFR mutations based on previous biopsy result and Cohort 2 will be patients with other cancer(s) suggested to have sensitivity to CPO301 in Part A.
* At least 1 measurable target lesion present and documented by CT or MRI according to RECIST v1.1
* ECOG performance status 0 or 1 at screening
* Life expectancy >12 weeks

Major Exclusion Criteria:

* Known, active, or uncontrolled central nervous system (CNS) metastasis or carcinomatous meningitis.
* Has AEs due to previous anti-tumor treatments not recovered to ≤Grade 1 (except for alopecia; some tolerable chronic toxicities of Grade 2 may be excluded after consultation with the sponsor, as judged by the investigator) according to NCI-CTCAE v5.0.
* Any serious and/or uncontrolled concurrent illness that may interfere with study participation

Prior therapy

* Received other investigational drugs or treatments within 4 weeks before the first dose of the investigational drug in the study
* The time interval between the latest anti-tumor treatment and the first dose of the investigational drug meets the following requirements: Have received anti-tumor treatments such as chemotherapy, radiotherapy, targeted therapy, immunotherapy and other clinical investigational drugs within 4 weeks before the first dose of the investigational drug; have received oral fluoropyrimidines, small molecule targeted drugs within 2 weeks before the first dose of the investigational drug; have received palliative radiotherapy or local therapy within 2 weeks before the first dose of investigational drug.
* Had major surgery within 4 weeks before the first dose of the investigational drug in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-06-13 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
To determine the dose to be used in Part B (RP2D) | through study completion, an average of 1 year
  To determine the recommended dose of CPO301 to be used as monotherapy in Part B (RP2D)
Safety and tolerability at RP2D of CPO301 as monotherapy | through study completion, an average of 1 year
  as measured by Incidence and severity of AEs per CTCAEv5.0

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | through study completion, an average of 1 year
  The pharmacokinetics (PK) profile of CPO301 will be assessed by measuring the blood concentration of the drug in the plasma at various timepoints and calculation of parameters, such as Peak Plasma Concentration (Cmax)
Expression of anti-drug antibody (ADA) | through study completion, an average of 1 year
  The expression of anti-drug antibodies (ADAs) following administration will be assessed by analysis of serum samples.
Efficacy assessment | through study completion, an average of 1 year
  To document any early indication of clinical efficacy

OTHER OUTCOMES:
Parts A and B, Exploratory: Correlatives | through study completion, an average of 1 year
  To explore the correlation between EGFR status (different mutations, or amplification levels) and efficacy in patients with advanced solid tumors and biomarkers relevant to CPO301 efficacy

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - Sarah Cannon Research Institute (SCRI) at HealthONE, Denver, Colorado
  - AdventHealth Cancer Institute, Celebration, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - NEXT Virginia, Fairfax, Virginia
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Cancer Centre - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No